CLINICAL TRIAL: NCT04765553
Title: A Randomized, Double-blinded, Placebo-controlled, Single Center, Phase I Study to Evaluate Pharmacokinetics, Pharmacodynamics and Safety of Emapalumab After a Single Intravenous Dose in Japanese Healthy Volunteers.
Brief Title: A Study to Evaluate Emapalumab in Japanese Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Sobi.emapalumab-102
Record Dates: First submitted 2021-01-18; First posted 2021-02-21 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Rare Diseases
MeSH Terms: conditions — Rare Diseases | interventions — Emapalumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- emapalumab (Active Comparator): emapalumab i.v infusion
  Interventions: Drug: NI-0501
- Placebo (Placebo Comparator): Saline i.v. infusion
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: NI-0501 — emapalumab single i.v infusion (1 mg/kg)
  Other Names: Gamifant
  Arms: emapalumab
Drug: Saline — Saline single i.v infusion
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, placebo controlled and double-blinded study to evaluate the pharmacokinetics (PK), pharmacodynamics (PD) and safety of a single dose (1 mg/kg) of emapalumab in adult healthy Japanese subjects.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled and double-blinded study to evaluate the PK, PD and safety of a single dose (1 mg/kg) of emapalumab in adult healthy Japanese subjects, performed in Japan. The subjects, 8 in total, will be randomized to receive either emapalumab or matching placebo in a 3:1 ratio (emapalumab: placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Japanese (male and female) subjects between 20 and 50 years (inclusive).
2. Body weight greater than 45 kg (female) or 50 kg (male) and a body mass index (BMI) >18 kg/m2 and < 30 kg/m2 (BMI= weight (kg) / height (m)²)
3. Vital signs in the following range:

   * Axillary body temperature: 35.2 - 37.5℃
   * Heart rate (after at least 3 minutes of rest, measured in the supine position): 40-100 bpm
   * BP < 140/80, mean of 3 readings after 15 minutes rest
4. Haemoglobin level equal or above 11 g/dL in females and 13 g/dL in males.
5. Subject having C-reactive protein (CRP) levels within the normal range (local laboratory range).
6. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant having agreed to use highly effective methods of contraception during dosing and for 6 months after receiving IMP.

   Highly effective contraception methods include:
   * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   * Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient, otherwise highly effective methods to be applied.
   * Use of oral (estrogen and progesterone) hormonal method of contraception, or placement of an intrauterine device (IUD) or intrauterine system (IUS)
   * In case of use of oral contraception women should have been stable on the same brand (or generic equivalent) for a minimum of 3 months before taking study treatment.

   Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago.
7. Signed informed consent.

Exclusion Criteria:

1. Any clinically significant abnormality in the results of the safety laboratory tests. Subjects presenting a minor deviation from laboratory ranges could be enrolled if the investigator judge it to be non-clinically significant
2. Any clinically significant abnormality on the screening electrocardiogram (ECG), as judged by the investigator
3. History or clinical evidence of any disease and/or existence of any surgical or medical condition that might interfere with the absorption, distribution, metabolism or excretion of the study drugs
4. Actual presence or occurrence of any bacterial, viral, parasitic or fungal infection within the 4 weeks preceding IMP infusion
5. Positive results from serology examination for Hepatitis B surface antigen (HBsAg), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV), syphilis (TP-antigen and RPR) or pregnancy
6. Positive stool test for Shigella or salmonella infection.
7. Positive results from Sars-CoV-2 screening within 96 hours prior to randomization
8. History or clinical evidence suggestive of active or latent tuberculosis at screening. (i.e. test positive to the interferon gamma (IFNγ)-release assay)
9. History or presence of any severe allergic reactions
10. History of hypersensitivity or allergy to any component of emapalumab and/or valaciclovir hydrochloride
11. History or presence of any malignancy
12. History or presence of drug or alcohol abuse
13. Subject with a smoking history within the last 6 months prior to the time of screening
14. Immunization with a live vaccine within 6 weeks prior to receiving IMP and 12 weeks after IMP infusion
15. Experience of collected blood corresponding to any of the following

    * Component blood donation within 2 weeks before the screening test and within 2 weeks before the first study drug administration
    * Collection of 200 mL or more of blood (blood donation, etc.) from 4 weeks before the screening test until admission
    * Male subject who has experience of collection of 400 mL or more of blood (blood donation, etc.) from 12weeks before the screening test until admission.
    * Female subject who has experience of collection of 400 mL or more of blood (blood donation, etc.) from 16weeks before the screening test until admission.
16. Usage of any prescription drugs within 2 weeks or over-the-counter medication including herbal supplements (with the exception of multi-vitamins) within 1 week before IMP administration without prior approval from the investigator
17. Positive pregnancy test at screening or Day -1
18. Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol
19. Enrollment in another concurrent clinical interventional study, or intake of another IMP, within four months or 5 half-lives (of the other IMP) prior to inclusion in this study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Furihata, MD, PhD, Principal Investigator — P-One Clinic, 4F, View Tower Hachioji, 8-1, Yokamachi, Hachioji-shi, Tokyo 192-0071, Japan
Locations (1):
- P-One Clinic, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Emapalumab | Placebo
Started | 6 | 2
Completed | 6 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emapalumab | Placebo | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Continuous [Median (Full Range); unit: years] | 35.0 [31 to 43] | 45 [44 to 46] | 40 [31 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Observed Concentration of Emapalumab
Description: The maximum observed concentration of emapalumab (Cmax)
Time Frame: Day 1 preinfusion, 1hr, 2hrs, 4hrs, 8hrs, 10hrs post dose, day 2, 3, 5, 8, week 2, 4, 6, 8, 10, 12, study completion week 14 or Withdrawal
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Emapalumab
Number analyzed (Participants) | 6
ng/mL | 23980 [22000 to 30600]

2. Primary Outcome: The Time at Which the Maximum Concentration of Emapalumab is Observed
Description: The time at which the maximum concentration of emapalumab is observed (Tmax)
Time Frame: Day 1 preinfusion, 1hr, 2 hrs, 4hrs, 8hrs, 10hrs, Day 2, 3, 5, 8, Week 2, 4, 6, 8, 10, 12, study completion week 14 or at Withdrawal
Measure: Median (Full Range); unit: Hours
Arm/Group | Emapalumab
Number analyzed (Participants) | 6
Hours | 2.000 [2.00 to 2.00]

3. Primary Outcome: Concentration of Emapalumab at End of Infusion
Description: Concentration of emapalumab at end of infusion (CEnd of inf))
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Emapalumab
Number analyzed (Participants) | 6
ng/mL | 23230 [21800 to 26800]

4. Primary Outcome: Area Under the Plasma Concentration-time Curve
Description: Area under the plasma concentration-time curve from emapalumab injection to time of last measurable concentration (AUClast)
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Emapalumab
Number analyzed (Participants) | 6
ng*h/mL | 11690000 [10300000 to 13400000]

5. Primary Outcome: Area Under the Concentration-time Curve Extrapolated to Infinity
Description: Area under the plasma concentration-time curve from emapalumab injection extrapolated to infinity (AUCinf)
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Emapalumab
Number analyzed (Participants) | 6
ng*h/mL | 12430000 [10800000 to 14600000]

6. Primary Outcome: Emapalumab Elimination Half-life
Description: Emapalumab elimination half-life (t1/2)
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Emapalumab
Number analyzed (Participants) | 6
Hours | 634.9 [489 to 683]

7. Primary Outcome: Apparent Total Body Clearance of Emapalumab From Plasma
Description: Apparent total body clearance of emapalumab from plasma (CL)
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: L/h
Arm/Group | Emapalumab
Number analyzed (Participants) | 6
L/h | 0.006136 [0.00395 to 0.00732]

8. Primary Outcome: Steady State Volume of Distribution
Description: Apparent volume of distribution at steady state (Vss)
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: L
Arm/Group | Emapalumab
Number analyzed (Participants) | 6
L | 4.953 [3.66 to 5.38]

9. Secondary Outcome: Overall Summary of Adverse Events
Description: Total number of reported adverse events
Time Frame: Continuously from start of emapalumab infusion up to 14 weeks
Measure: Number; unit: number of events
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
number of events
  All Treatment emergent adverse events (TEAEs) | 3 | 1
  Adverse Drug Reactions (ADRs) | 3 | 0
  Serious TEAEs | 0 | 0
  Serious ADRs | 0 | 0
  TEAEs leading to drug withdrawn | 0 | 0
  ADRs leading to drug withdrawn | 0 | 0
  TEAEs leading to dose reduced | 0 | 0
  ADRs leading to dose reduced | 0 | 0
  TEAEs leading to drug interrupted | 0 | 0
  ADRs leading to drug interrupted | 0 | 0
  TEAEs leading to death | 0 | 0
  ADRs leading to death | 0 | 0
  Infusion Related Reactions, (IRRs) | 2 | 0

10. Secondary Outcome: Change in Levels of Aspartate Aminotransferase
Description: Change from baseline in levels of Aspartate aminotransferase (AST)
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples.
Measure: Median (Full Range); unit: IU/L
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
IU/L
  Day 1 | 0.5 [-4 to 2] | 2.5 [0 to 5]
  Day 2 | -0.5 [-5 to 1] | 5.0 [-1 to 11]
  Day 3 | -2.5 [-7 to 0] | 1.5 [-4 to 7]
  Day 5 | -1.5 [-5 to 1] | 9.0 [-4 to 22]
  Day 8 | 1.0 [-3 to 9] | 11.5 [-1 to 24]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -2 [-5 to 1] | 7.0 [7 to 7]
  Week 4 | -0.5 [-4 to 18] | 6.5 [6 to 7]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -2.0 [-5 to 2] | 0.5 [0 to 1]
  Week 10 | -1.5 [-3 to 4] | 6.5 [4 to 9]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -2.0 [-6 to 8] | 5.0 [0 to 10]

11. Secondary Outcome: Change in Levels of Alanine Aminotransferase
Description: Change from baseline in levels of Alanine aminotransferase (ALT)
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: IU/L
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
IU/L
  Day 1 | 0.5 [-4 to 5] | 1.0 [-1 to 3]
  Day 2 | 0.0 [-5 to 4] | 2.5 [-2 to 7]
  Day 3 | -2.0 [-7 to 0] | 0.5 [-6 to 7]
  Day 5 | -0.5 [-4 to 5] | 12.0 [-7 to 31]
  Day 8 | 4.5 [-5 to 19] | 18.5 [-6 to 43]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -3.0 [-11 to 4] | 15.0 [15 to 15]
  Week 4 | 1.0 [-8 to 12] | 19.5 [10 to 29]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -4.0 [-7 to 6] | 0.0 [-3 to 3]
  Week10 | 2.0 [-5 to 8] | 8.5 [7 to 10]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 0.0 [-9 to 17] | 5.5 [-1 to 12]

12. Secondary Outcome: Change in Levels of Direct Bilirubin
Description: Change from baseline in levels of Direct Bilirubin
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | 0.15 [0.0 to 0.3] | 0.05 [0.0 to 0.1]
  Day 2 | 0.15 [0.0 to 0.5] | 0.00 [-0.1 to 0.1]
  Day 3 | 0.10 [-0.1 to 0.2] | -0.05 [-0.1 to 0.0]
  Day 5 | 0.05 [-0.1 to 0.1] | -0.05 [-0.1 to 0.0]
  Day 8 | 0.10 [-0.1 to 0.1] | 0.00 [0.0 to 0.0]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | 0.00 [-0.1 to 0.1] | -0.10 [-0.1 to -0.1]
  Week 4 | 0.05 [0.0 to 0.1] | 0.00 [0.0 to 0.0]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | 0.10 [-0.1 to 0.1] | 0.00 [0.0 to 0.0]
  Week 10 | 0.05 [0.0 to 0.2] | -0.05 [-0.1 to 0.0]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 0.00 [0.0 to 0.1] | -0.05 [-0.1 to 0.0]

13. Secondary Outcome: Change in Levels of Total Bilirubin
Description: Change from baseline in levels of Total Bilirubin
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | 0.35 [0.1 to 1.3] | 0.30 [0.2 to 0.4]
  Day 2 | 0.55 [0.0 to 1.7] | 0.10 [-0.1 to 0.3]
  Day 3 | 0.15 [-0.5 to 0.8] | -0.10 [-0.3 to 0.1]
  Day 5 | 0.10 [-0.4 to 0.4] | -0.20 [-0.3 to -0.1]
  Day 8 | 0.20 [-0.5 to 0.6] | 0.05 [-0.1 to 0.2]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -0.05 [-0.5 to 0.2] | -0.20 [-0.2 to -0.2]
  Week 4 | 0.15 [-0.3 to 0.5] | -0.05 [-0.1 to 0.0]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | 0.10 [-0.4 to 0.5] | 0.05 [-0.1 to 0.2]
  Week 10 | 0.15 [-0.2 to 0.6] | 0.00 [-0.1 to 0.1]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 0.10 [-0.3 to 0.2] | -0.15 [-0.5 to 0.2]

14. Secondary Outcome: Change in Levels of Uric Acid
Description: Change from baseline in levels of Uric acid
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | 0.15 [-0.2 to 0.6] | 0.10 [-0.1 to 0.3]
  Day 2 | 0.40 [0.1 to 0.8] | 0.15 [-0.3 to 0.6]
  Day 3 | 0.40 [-0.1 to 0.8] | 0.15 [-0.4 to 0.7]
  Day 5 | 0.35 [-0.1 to 1.6] | 0.20 [-0.2 to 0.6]
  Day 8 | 0.25 [-0.4 to 1.2] | 0.20 [0.0 to 0.4]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -0.10 [-0.6 to 1.1] | -0.40 [-0.4 to -0.4]
  Week 4 | 0.25 [-0.6 to 0.5] | -0.05 [-0.5 to 0.4]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | 0.00 [-0.6 to 0.7] | 0.10 [-0.2 to 0.4]
  Week 10 | 0.40 [-0.2 to 2.2] | 0.55 [0.3 to 0.8]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 0.10 [-0.7 to 0.5] | 0.85 [0.3 to 1.4]

15. Secondary Outcome: Change in Levels of Alkaline Phosphatase
Description: Change from baseline in levels of Alkaline phosphatase
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: U/L
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
U/L
  Day 1 | -34.0 [-45 to 13] | 16.0 [15 to 17]
  Day 2 | -26.5 [-46 to 25] | 16.0 [13 to 19]
  Day 3 | -23.5 [-42 to 30] | 22.0 [10 to 34]
  Day 5 | -28.0 [-53 to 31] | 17.0 [4 to 30]
  Day 8 | -6.5 [-20 to 27] | 35.0 [22 to 48]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | 9.5 [-44 to 26] | 26.0 [26 to 26]
  Week 4 | 4.0 [-9 to 25] | 33.5 [17 to 50]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | 8.0 [-40 to 42] | 22.0 [19 to 25]
  Week 10 | -0.5 [-25 to 22] | 40.0 [19 to 61]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -15.0 [-51 to 45] | 33.0 [17 to 49]

16. Secondary Outcome: Change in Levels of Total Protein
Description: Change from baseline in levels of Total protein
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: g/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
g/dL
  Day 1 | 0.25 [-0.2 to 0.4] | 0.30 [0.2 to 0.4]
  Day 2 | 0.25 [-0.2 to 0.4] | 0.25 [0.2 to 0.3]
  Day 3 | 0.20 [-0.4 to 0.7] | 0.35 [0.2 to 0.5]
  Day 5 | 0.15 [-0.5 to 0.6] | 0.00 [-0.1 to 0.1]
  Day 8 | 0.50 [0.2 to 0.8] | 0.65 [0.4 to 0.9]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -0.05 [-0.2 to 0.4] | 0.10 [0.1 to 0.1]
  Week 4 | 0.05 [-0.4 to 0.6] | -0.10 [-0.4 to 0.2]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -0.10 [-0.4 to 0.2] | 0.05 [-0.4 to 0.5]
  Week 10 | 0.4 [0.3 to 0.7] | 0.15 [-0.1 to 0.4]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 0.10 [-0.2 to 0.4] | 0.55 [0.2 to 0.9]

17. Secondary Outcome: Change in Levels of Albumin
Description: Change from baseline in levels of Albumin
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: g/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
g/dL
  Day 1 | 0.10 [-0.2 to 0.2] | 0.35 [0.3 to 0.4]
  Day 2 | 0.05 [0.0 to 0.2] | 0.30 [0.3 to 0.3]
  Day 3 | -0.15 [-0.2 to 0.2] | 0.20 [0.1 to 0.3]
  Day 5 | 0.00 [-0.1 to 0.2] | 0.20 [0.2 to 0.2]
  Day 8 | 0.30 [0.2 to 0.6] | 0.45 [0.3 to 0.6]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -0.05 [-0.3 to 0.1] | 0.00 [0.0 to 0.0]
  Week 4 | 0.10 [-0.6 to 0.3] | 0.10 [-0.1 to 0.3]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -0.10 [-0.4 to 0.0] | 0.00 [-0.3 to 0.3]
  Week 10 | 0.30 [0.2 to 0.4] | 0.05 [-0.1 to 0.2]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 0.00 [-0.2 to 0.1] | 0.25 [0.0 to 0.5]

18. Secondary Outcome: Change in Levels of Prothrombin Time/International Normalized Ratio
Description: Change from baseline in levels of Prothrombin Time/International Normalized Ratio (PTINR)
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: Unitless
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
Unitless
  Day 1 | 0.065 [0.02 to 0.10] | -0.005 [-0.05 to 0.04]
  Day 2 | 0.045 [-0.05 to 0.10] | -0.035 [-0.08 to 0.01]
  Day 3 | 0.075 [0.00 to 0.11] | 0.010 [-0.05 to 0.07]
  Day 5 | 0.015 [-0.03 to 0.06] | -0.025 [-0.06 to 0.01]
  Day 8 | -0.005 [-0.03 to 0.08] | -0.055 [-0.10 to -0.01]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -0.020 [-0.07 to 0.07] | -0.060 [-0.06 to -0.06]
  Week 4 | -0.040 [-0.10 to 0.09] | -0.055 [-0.11 to 0.00]
  Week 6 | -0.050 [-0.09 to 0.07] | -0.050 [-0.09 to -0.01]
  Week 10 | -0.030 [-0.08 to 0.06] | -0.065 [-0.14 to 0.01]
  Week 14 | -0.030 [-0.05 to 0.05] | -0.085 [-0.17 to 0.00]

19. Secondary Outcome: Change in Levels of Fibrinogen
Description: Change from baseline in levels of Fibrinogen
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | 6.0 [-48 to 18] | 49.5 [40 to 59]
  Day 2 | 53.0 [-38 to 125] | 103.5 [92 to 115]
  Day 3 | 60.0 [-184 to 190] | -97.0 [-110 to -84]
  Day 5 | 75.5 [-7 to 174] | 6.0 [-38 to 50]
  Day 8 | 93.5 [-134 to 145] | 84.0 [53 to 115]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -5.5 [-135 to 78] | 2.5 [-5 to 10]
  Week 4 | -5.5 [-135 to 78] | 2.5 [-5 to 10]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -14.0 [-34 to 20] | 23.5 [-3 to 50]
  Week 10 | 10.5 [-6 to 102] | -5.0 [-19 to 9]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -43.0 [-122 to 86] | 7.5 [-9 to 24]

20. Secondary Outcome: Change in Levels of Complement C3
Description: Change from baseline in levels of Complement C3
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | 4.0 [-2 to 13] | 11.5 [8 to 15]
  Day 2 | 3.5 [-1 to 16] | 4.5 [3 to 6]
  Day 3 | 12.5 [-3 to 30] | 9.0 [5 to 13]
  Day 5 | 14.5 [-4 to 40] | 3.0 [0 to 6]
  Day 8 | 20.0 [4 to 32] | 16.5 [8 to 25]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | 10.5 [0 to 18] | 3.0 [3 to 3]
  Week 4 | 0.5 [-8 to 17] | 3.0 [-1 to 7]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -1.0 [-8 to 8] | -0.5 [-7 to 6]
  Week 10 | 6.5 [2 to 20] | 4.5 [-1 to 10]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -9.0 [-15 to 14] | 5.5 [-5 to 16]

21. Secondary Outcome: Change in Levels of Creatinine
Description: Change from baseline in levels of Creatinine
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | 0.030 [-0.03 to 0.08] | 0.095 [0.05 to 0.14]
  Day 2 | 0.010 [0.01 to 0.02] | 0.020 [-0.04 to 0.08]
  Day 3 | 0.010 [-0.04 to 0.05] | 0.025 [-0.05 to 0.10]
  Day 5 | 0.055 [-0.02 to 0.07] | 0.035 [0.00 to 0.07]
  Day 8 | -0.005 [-0.03 to 0.04] | -0.005 [-0.04 to 0.03]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -0.035 [-0.09 to 0.14] | -0.060 [-0.06 to -0.06]
  Week 4 | -0.040 [-0.12 to 0.07] | 0.025 [-0.01 to 0.06]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -0.030 [-0.11 to 0.17] | 0.010 [-0.07 to 0.09]
  Week 10 | -0.020 [-0.10 to 0.13] | -0.010 [-0.07 to 0.05]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 0.010 [-0.13 to 0.12] | 0.125 [0.03 to 0.22]

22. Secondary Outcome: Change in Levels of C-reactive Protein
Description: Change from baseline in levels of C-reactive protein (CRP)
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | 0.000 [-0.03 to 0.05] | -0.015 [-0.05 to 0.02]
  Day 2 | 0.105 [-0.01 to 0.94] | 0.030 [-0.08 to 0.14]
  Day 3 | 0.645 [-0.01 to 2.28] | 0.025 [-0.09 to 0.14]
  Day 5 | 0.155 [-0.01 to 0.54] | -0.035 [-0.08 to 0.01]
  Day 8 | 0.050 [0.00 to 0.13] | -0.025 [-0.08 to 0.03]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | 0.010 [-0.02 to 0.04] | -0.050 [-0.05 to -0.05]
  Week 4 | 0.000 [-0.04 to 0.36] | 0.065 [0.00 to 0.13]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | 0.030 [-0.02 to 0.07] | -0.060 [-0.10 to -0.02]
  Week10 | 0.005 [-0.06 to 0.07] | -0.025 [-0.08 to 0.03]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -0.010 [-0.01 to 0.10] | -0.025 [-0.09 to 0.04]

23. Secondary Outcome: Change in Levels of Sodium
Description: Change from baseline in levels of Sodium
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mEq/L
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mEq/L
  Day 1 | -1.0 [-4 to 2] | 3.5 [3 to 4]
  Day 2 | -0.5 [-2 to 1] | 1.5 [1 to 2]
  Day 3 | -1.5 [-3 to 0] | 2.0 [2 to 2]
  Day 5 | 0.00 [-4 to 1] | 2.5 [2 to 3]
  Day 8 | 0.0 [-4 to 2] | 2.0 [2 to 2]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -0.5 [-3 to 3] | 1.0 [1 to 1]
  Week 4 | -0.5 [-6 to 3] | 3.5 [3 to 4]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | 0.0 [-3 to 2] | 5.0 [3 to 7]
  Week 10 | -1.5 [-5 to 2] | 0.5 [0 to 1]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -1.0 [-2 to 2] | 3.5 [0 to 7]

24. Secondary Outcome: Change in Levels of Potassium
Description: Change from baseline in levels of Potassium
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mEq/L
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mEq/L
  Day 1 | 0.00 [-0.5 to 0.2] | 0.60 [0.5 to 0.7]
  Day 2 | 0.00 [-0.8 to 0.4] | 0.15 [0.0 to 0.3]
  Day 3 | 0.15 [-0.5 to 0.3] | 0.40 [0.0 to 0.8]
  Day 5 | 0.15 [0.1 to 0.4] | 0.00 [-0.1 to 0.1]
  Day 8 | -0.15 [-0.6 to 0.2] | -0.25 [-0.4 to -0.1]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | 0.15 [-0.2 to 0.3] | 0.10 [0.1 to 0.1]
  Week 4 | 0.00 [-0.2 to 0.3] | 0.35 [0.2 to 0.5]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | 0.00 [-0.1 to 0.1] | 0.40 [0.1 to 0.7]
  Week 10 | 0.05 [-0.4 to 0.5] | -0.20 [-0.3 to -0.1]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 0.00 [-0.02 to 0.3] | 0.30 [0.0 to 0.6]

25. Secondary Outcome: Change in Levels of Calcium
Description: Change from baseline in levels of Calcium
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | -0.05 [-0.8 to 0.2] | 0.40 [0.3 to 0.5]
  Day 2 | 0.00 [-0.6 to 0.3] | 0.15 [0.1 to 0.2]
  Day 3 | -0.10 [-0.6 to 0.7] | 0.30 [0.2 to 0.4]
  Day 5 | 0.05 [-0.5 to 0.5] | 0.20 [0.1 to 0.3]
  Day 8 | 0.15 [-0.1 to 0.4] | 0.10 [-0.1 to 0.3]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -0.05 [-0.6 to 0.4] | 0.10 [0.1 to 0.1]
  Week 4 | -0.15 [-0.9 to 0.3] | -0.05 [-0.1 to 0.0]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -0.40 [-1.0 to 0.5] | 0.15 [-0.4 to 0.7]
  Week 10 | 0.30 [0.0 to 0.6] | 0.00 [-0.1 to 0.1]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 0.00 [-0.3 to 0.5] | 0.55 [0.2 to 0.9]

26. Secondary Outcome: Change in Levels of Glucose
Description: Change from baseline in levels of Glucose
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | -9.0 [-13 to 0] | -3.0 [-5 to -1]
  Day 2 | -1.0 [-5 to 4] | 0.5 [-1 to 2]
  Day 3 | 0.5 [-6 to 6] | 3.0 [0 to 6]
  Day 5 | -4.5 [-7 to 0] | -2.0 [-5 to 1]
  Day 8 | -7.5 [-14 to -4] | 0.0 [-3 to 3]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -2.0 [-11 to 0] | 2.0 [2 to 2]
  Week 4 | -1.0 [-6 to 10] | 3.0 [0 to 6]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | 0.0 [0 to 5] | 4.5 [4 to 5]
  Week 10 | 1.5 [-4 to 4] | 0.5 [-1 to 2]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 1.0 [-5 to 9] | 0.5 [-2 to 3]

27. Secondary Outcome: Change in Levels of HDL
Description: Change from baseline in levels of HDL
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | -2.0 [-8 to 3] | 0.0 [0 to 0]
  Day 2 | -3.5 [-8 to 0] | -1.0 [-2 to 0]
  Day 3 | -4.0 [-11 to 0] | 1.0 [-1 to 3]
  Day 5 | -8.0 [-14 to -2] | -1.5 [-4 to 1]
  Day 8 | -7.5 [-14 to -2] | 2.5 [0 to 5]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -7.0 [-9 to 2] | 0.0 [0 to 0]
  Week 4 | -2.0 [-8 to 11] | -2.0 [-5 to 1]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -5.0 [-7 to 6] | -1.0 [-2 to 0]
  Week 10 | 0.5 [-4 to 6] | -0.5 [-3 to 2]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -5.0 [-10 to -2] | 0.5 [-2 to 3]

28. Secondary Outcome: Change in Levels of LDL
Description: Change from baseline in levels of LDL
Time Frame: Baselilne, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | 11.0 [-5 to 13] | 16.5 [15 to 18]
  Day 2 | 5.5 [-13 to 17] | 17.0 [13 to 21]
  Day 3 | 3.5 [-32 to 23] | 19.5 [14 to 25]
  Day 5 | 3.0 [-40 to 15] | 7.5 [5 to 10]
  Day 8 | 7.0 [-25 to 22] | 13.0 [1 to 25]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -7.0 [-25 to 19] | 17.0 [17 to 17]
  Week 4 | 2.0 [-22 to 19] | 0.0 [-7 to 7]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | 3.0 [-24 to 39] | 3.5 [-3 to 10]
  Week 10 | 9.0 [-2 to 32] | 3.5 [-15 to 22]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -8.0 [-11 to 8] | 19.5 [7 to 32]

29. Secondary Outcome: Change in Levels of BUN/Urea Haematology
Description: Change from baseline in levels of BUN/Urea haematology
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | -1.35 [-3.6 to 0.0] | -1.60 [-2.1 to -1.1]
  Day 2 | -0.55 [-2.8 to 1.7] | 2.55 [0.9 to 4.2]
  Day 3 | -1.05 [-2.2 to -0.4] | 1.30 [-1.1 to 3.7]
  Day 5 | 0.80 [-1.7 to 1.6] | 2.00 [0.3 to 3.7]
  Day 8 | -2.05 [-5.3 to 2.3] | -1.50 [-3.0 to 0.0]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -1.90 [-2.6 to 2.8] | -2.30 [-2.3 to -2.3]
  Week 4 | -1.40 [-6.6 to 4.4] | 3.10 [0.8 to 5.4]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -2.20 [-4.4 to 4.9] | -1.25 [-2.7 to 0.2]
  Week 10 | 0.95 [-6.2 to 2.4] | -1.15 [-4.8 to 2.5]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -1.70 [-2.7 to -1.4] | 2.75 [-0.9 to 6.4]

30. Secondary Outcome: Change in Levels of Hemoglobin
Description: Change from baseline in levels of Hemoglobin
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: g/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
g/dL
  Day 1 | 0.4 [-0.6 to 0.6] | 0.75 [0.6 to 0.9]
  Day 2 | 0.35 [-0.2 to 0.8] | 0.55 [0.3 to 0.8]
  Day 3 | 0.20 [-0.5 to 0.7] | 0.45 [0.0 to 0.9]
  Day 5 | 0.25 [-0.4 to 1.1] | 0.25 [0.1 to 0.4]
  Day 8 | 0.75 [0.5 to 0.9] | 0.7 [0.4 to 1.0]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -0.25 [-0.7 to 0.7] | 0.10 [0.1 to 0.1]
  Week 4 | 0.00 [-0.9 to 0.8] | 0.20 [-0.2 to 0.6]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -0.20 [-0.6 to 0.5] | 0.05 [-0.5 to 0.6]
  Week 10 | 0.90 [0.3 to 1.5] | 0.65 [0.5 to 0.8]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 0.20 [-0.4 to 0.7] | 1.25 [1.2 to 1.3]

31. Secondary Outcome: Change in Levels of Hematocrit
Description: Change from baseline in levels of Hematocrit
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: % of red blood cells in blood
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
% of red blood cells in blood
  Day 1 | 1.6 [-1.6 to 2.8] | 2.80 [2.3 to 3.3]
  Day 2 | 1.10 [-0.3 to 3.0] | 2.10 [1.5 to 2.7]
  Day 3 | 0.70 [-1.3 to 2.9] | 1.55 [0.7 to 2.4]
  Day 5 | 0.90 [-1.2 to 3.6] | 0.7 [0.2 to 1.2]
  Day 8 | 2.70 [1.7 to 3.5] | 2.15 [1.3 to 3.0]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -0.40 [-1.9 to 4.2] | 0.3 [0.3 to 0.3]
  Week 4 | 0.15 [-2.2 to 2.6] | 0.95 [-0.1 to 2.0]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | 1.00 [-1.1 to 1.9] | 0.85 [-1.6 to 3.3]
  Week 10 | 3.05 [1.2 to 4.0] | 2.70 [2.1 to 3.3]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 0.1 [-1.4 to 1.4] | 2.45 [2.4 to 2.5]

32. Secondary Outcome: Change in Levels of Platelet Count
Description: Change from baseline in levels of Platelet count
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: x10^10/L
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
x10^10/L
  Day 1 | 0.40 [0.2 to 1.2] | 1.20 [1.1 to 1.3]
  Day 2 | -0.15 [-1.3 to 0.9] | 1.10 [0.9 to 1.3]
  Day 3 | -0.1 [-2.3 to 0.3] | 1.40 [1.4 to 1.4]
  Day 5 | 0.05 [-0.4 to 1.6] | 1.8 [1.6 to 2.0]
  Day 8 | 1.8 [0.3 to 5.7] | 3.70 [3.2 to 4.2]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | 0.70 [-0.6 to 3.1] | 2.30 [2.3 to 2.3]
  Week 4 | 0.05 [-0.2 to 3.3] | 1.55 [0.7 to 2.4]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | 0.4 [-2.7 to 1.6] | 3.10 [2.8 to 3.4]
  Week 10 | 0.5 [-0.5 to 4.0] | 2.40 [1.6 to 3.2]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -0.10 [-3.2 to 1.7] | 4.65 [4.1 to 5.2]

33. Secondary Outcome: Change in Levels of Neutrophils
Description: Change from baseline in levels of Neutrophils
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: % of white blood cells
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
% of white blood cells
  Day 1 | -0.30 [-4.5 to 3.6] | 0.35 [-7.5 to 8.2]
  Day 2 | 17.45 [-0.5 to 21.1] | -0.40 [-6.0 to 5.2]
  Day 3 | 9.70 [-1.1 to 12.2] | -0.85 [-3.0 to 1.3]
  Day 5 | 0.75 [-6.4 to 9.2] | -16.25 [-30.8 to -1.7]
  Day 8 | 1.65 [-4.0 to 6.8] | 1.30 [0.7 to 1.9]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | 2.50 [-2.1 to 17.9] | 5.10 [5.1 to 5.1]
  Week 4 | -1.05 [-4.1 to 7.4] | 2.10 [-1.6 to 5.8]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -4.10 [-9.5 to 8.3] | 0.55 [-1.9 to 3.0]
  Week 10 | 1.45 [-9.7 to 8.6] | 0.95 [-1.4 to 3.3]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -5.40 [-10.5 to 1.7] | 1.65 [-4.7 to 8.0]

34. Secondary Outcome: Change in Levels of Red Blood Cells
Description: Change from baseline in levels of Red blood cells
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: cellsx10^10/L
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
cellsx10^10/L
  Day 1 | 18 [-20 to 30] | 27.0 [25 to 29]
  Day 2 | 13.5 [-7 to 29] | 20.0 [13 to 27]
  Day 3 | 9.0 [-15 to 33] | 15.0 [6 to 24]
  Day 5 | 12.0 [-14 to 43] | 8.5 [3 to 14]
  Day 8 | 29.5 [21 to 33] | 23.5 [14 to 33]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -4.0 [-24 to 27] | 0.0 [0 to 0]
  Week 4 | -1.0 [-27 to 24] | 2.0 [-9 to 13]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -6.0 [-23 to 11] | -0.5 [-23 to 22]
  Week 10 | 23.0 [-1 to 32] | 20.0 [13 to 27]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -6.0 [-25 to -2] | 18.5 [16 to 21]

35. Secondary Outcome: Change in Levels of Immunoglobulin Levels
Description: Change from baseline in levels of Immunoglobulin levels (IgG)
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | 69.5 [-60 to 100] | 119.5 [119 to 120]
  Day 2 | 28.5 [7 to 78] | 72.0 [66 to 78]
  Day 3 | 5.0 [-41 to 67] | 78 [62 to 94]
  Day 5 | 6.0 [-79 to 92] | 16.0 [5 to 27]
  Day 8 | 125.5 [105 to 148] | 156.5 [76 to 237]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | 14.5 [-52 to 105] | 48.0 [48 to 48]
  Week 4 | 29.5 [-63 to 182] | 34.5 [1 to 68]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | 2.0 [-82 to 135] | 36.0 [-40 to 112]
  Week 10 | 98.0 [37 to 267] | 49.5 [-14 to 113]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | 1.0 [-99 to 185] | 89.5 [-24 to 203]

36. Secondary Outcome: Change in Levels of Coagulation Profile
Description: Change from baseline in Activated Partial Thromboplastin Clotting Time (APTT)
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of patients analyzed are the number of available samples.
Measure: Median (Full Range); unit: sec
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
sec
  Day 1 | 0.85 [0.4 to 2.1] | 0.4 [0.2 to 0.6]
  Day 2 | -0.30 [-1.2 to 2.6] | -0.65 [-0.9 to -0.4]
  Day 3 | 0.4 [-0.9 to 2.2] | 1.80 [1.2 to 2.4]
  Day 5 | -1.40 [-2.0 to 2.1] | -0.80 [-1.4 to -0.2]
  Day 8 | 1.40 [-0.8 to 3.5] | 0.30 [0.0 to 0.6]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | -0.55 [-1.5 to 2.1] | 0.5 [0.5 to 0.5]
  Week 4 | -0.15 [-2.0 to 2.8] | -2.25 [-2.3 to -2.2]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -0.90 [-2.4 to 1.3] | -0.50 [-1.3 to 0.3]
  Week 10 | 1.50 [-1.9 to 3.8] | -2.60 [-3.5 to -1.7]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -1.80 [-3.1 to 3.5] | -1.25 [-3.4 to 0.9]

37. Secondary Outcome: Presence of Anti-drug Antibodies and Neutralizing Antibodies
Description: Presence of anti-drug antibodies (ADA) and neutralizing antibodies (nAb)
Time Frame: From Day 1 to Week 14
Population: Number of analyzed are the number of available samples
Measure: Count of Participants; unit: Participants
Arm/Group | Emapalumab
Number analyzed (Participants) | 6
Participants
  Baseline | 0
  Week 14: number analyzed (Participants) | 5
  Week 14 | 0

38. Secondary Outcome: Change in Levels of Complement C4
Description: Change from baseline in levels of Complement C4
Time Frame: Baseline, Days 1,2,3,5,8, Weeks 2,4,6,10, and Study Completion Visit (Week 14)
Population: Number of analyzed are the number of available samples
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Emapalumab | Placebo
Number analyzed (Participants) | 6 | 2
mg/dL
  Day 1 | 0.0 [-1 to 2] | 2.5 [2 to 3]
  Day 2 | 1.0 [-1 to 4] | 2.0 [1 to 3]
  Day 3 | 3.0 [-1 to 8] | 3.0 [1 to 5]
  Day 5 | 4.5 [-1 to 12] | 2.5 [0 to 5]
  Day 8 | 6.0 [1 to 11] | 6.0 [3 to 9]
  Week 2: number analyzed (Participants) | 6 | 1
  Week 2 | 2.0 [1 to 4] | 4.0 [4 to 4]
  Week 4 | 0.0 [-4 to 3] | -1.0 [-3 to 1]
  Week 6: number analyzed (Participants) | 5 | 2
  Week 6 | -1.0 [-2 to 3] | 1.5 [-2 to 5]
  Week 10 | -1.5 [-3 to 0] | -1.5 [-3 to 0]
  Week 14: number analyzed (Participants) | 5 | 2
  Week 14 | -4.0 [-7 to 6] | 1.5 [-3 to 6]

39. Secondary Outcome: Presence of Neutralizing Antibodies
Description: Presence of neutralizing antibodies (nAb)
Time Frame: From Day 1 to Week 14
Measure: Count of Participants; unit: Participants
Arm/Group | Emapalumab
Number analyzed (Participants) | 6
Participants | NA — None of the subjects had positive anti-drug-antibody result, so this analyse was not done

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of dosing the IMP up to week 14
Arm/Group | Emapalumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 3/6 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emapalumab (N=6) | Placebo (N=2)
C-reactive protein increased (Investigations) | 3 (3) | 0 (0)
Feeling hot (General disorders) | 2 (2) | 0
Malaise (General disorders) | 2 (2) | 0
Pyrexia (General disorders) | 1 (1) | 0
Nasopharyngitis (Infections and infestations) | 1 (1) | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT04765553/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT04765553/SAP_001.pdf